CLINICAL TRIAL: NCT03560206
Title: Effects of Family Sodium Watcher Program on Outcomes in Heart Failure Patient-Family Caregiver Dyads
Acronym: FAMSWAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misook L. Chung (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Misook L. Chung, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 46045; R01NR012967 (NIH)
Record Dates: First submitted 2015-01-06; First posted 2018-06-18 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
Keywords: Diet, low-sodium; caregivers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: a randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family SWaP intervention (Experimental): an educational-behavioral intervention consisting of 6 weekly education sessions (45 minutes) followed by 5 bi-weekly sessions (15-20 minutes) that will be held at the dyad's preferred time delivered to their homes using a video conferencing program through a mini iPad.
  Interventions: Behavioral: Family SWaP intervention
- Usual Care (Active Comparator): The usual care group will receive their routine medical and nursing care for heart failure that consists of a recommendation to follow a sodium restricted diet without explicit skills training to do so.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Family SWaP intervention — The Family Sodium Watcher Program (Family SWaP) proposed in this study incorporates the use of a unique electronic salt monitoring device that easily measures salt content in food-the major source of sodium. The intervention is designed to improve adherence to a sodium restricted diet by both patients and family caregivers through education and strategies for gradual taste adaptation to low salt foods. The Family SWaP intervention (6 weekly 45-minute sessions followed by 5 bi-weekly booster sessions) will be delivered remotely using a video-conferencing program on an iPad tablet.
  Other Names: Family SWaP
  Arms: Family SWaP intervention
Behavioral: usual care — The usual care group will receive their routine medical and nursing care for heart failure that consists of a recommendation to follow a sodium restricted diet without explicit skills training to do so.
  Arms: Usual Care

SUMMARY:
The Family Sodium Watcher program in this study is designed to improve adherence to a sodium restricted diet in patients with HF using strategies that educate both patients and family caregivers about sodium monitoring and that stress a gradual progressive adaptation to low sodium food for both patients and family caregivers.

DETAILED DESCRIPTION:
Heart failure (HF) emerged as a significant public health threat in the 1990s and has now reached epidemic proportions. Despite advances in the medical treatment of HF, patients with HF face frequent hospitalizations for acute exacerbations. Inadequate self-care strategies, in particular non-adherence to a sodium restricted diet (SRD), is a main cause of these rehospitalizations. Prior interventions to increase adherence have focused on increasing knowledge about restricting sodium in the diet have met with limited success. Unaddressed by these interventions are the major barriers of measuring and tracking daily sodium intake, family members who continue to eat high sodium diets, and a preference for salty foods-particularly in the elderly who have a decreased sense of taste. It is possible to retrain the taste buds to enjoy low salt foods by gradually reducing the amount of sodium in foods over the course of 16 weeks. This retraining works best with direct involvement and support from family members. The Family Sodium Watcher Program (Family SWaP) proposed in this study incorporates the use of a unique electronic salt monitoring device that easily measures salt content in food-the major source of sodium. The intervention is designed to improve adherence to a SRD by both patients and family caregivers through education and strategies for gradual taste adaptation to low salt foods.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will:

* have diagnosis of chronic HF with either preserved or reduced ejection fraction
* have a dedicated primary family caregiver
* be able to speak and write English

Eligible caregivers will:

* be a primary caregiver identified by the patient
* the spouse, committed partner, or family member living with the HF patient
* be able to speak and understand English
* have no obvious major clinical cognitive impairment that would impair ability to give informed consent
* have no major co-morbidities (i.e. HF, cancer, renal/liver failure, or uncontrolled diabetes as determined by self-report).

Exclusion Criteria:

Patients will be excluded if they have:

* major clinical cognitive impairment (i.e., dementia, Alzheimer disease, and severe stroke)
* a co-existing terminal illness (e.g., cancer)
* a referral for heart transplantation
* a dietary prescription that prevents following a 2-3 gram sodium diet (e.g., clinician does not support use of a SRD).
* no dedicated caregivers

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misook L Chung, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky HealthCare, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited a total of 316 individuals consisting of 158 patients with heart failure and 158 primary caregivers at outpatient cardiology clinics in one academic medical center and one community medical center.
Pre-assignment Details: As a result of the screening of 5,365 patients, a total of 819 dyads who met the inclusion criteria and 214 dyads verbally agreed to participate (26.1% recruitment rate). Of these, 199 dyads provided written consent,but 41 dyads withdrew before the home visit for baseline data collection. Thus, only158 dyads (316 individuals: 158 patients and 158 caregivers) completed the baseline assessment. Thus, we reported the final sample of 158 patients with heart failure in this report.
Groups:
- Family SWaP Intervention: an educational-behavioral intervention consisting of 6 weekly education sessions (45 minutes) followed by 5 bi-weekly sessions (15-20 minutes) that will be held at the dyad's preferred time delivered to their homes using a video conferencing program through a mini iPad.
  Family SWaP intervention with mini iPad: The Family Sodium Watcher Program (Family SWaP) proposed in this study incorporates the use of a unique electronic salt monitoring device that easily measures salt content in food-the major source of sodium. The intervention is designed to improve adherence to a sodium restricted diet by both patients and family caregivers through education and strategies for gradual taste adaptation to low salt foods. The Family SWaP intervention (6 weekly 45-minute sessions followed by 5 bi-weekly booster sessions) will be delivered remotely using a video-conferencing program on an iPad tablet.
Period: Overall Study
Arm/Group | Family SWaP Intervention | Usual Care
Started | 158 | 158
Completed | 108 | 140
Not Completed | 50 | 18
Not completed — Lost to Follow-up | 19 | 11
Not completed — Withdrawal by Subject | 2 | 4
Not completed — caregivers' health condition and not becoming non-caregiver | 5 | 0
Not completed — Busy schedule | 14 | 2
Not completed — patients' new health condition such as cancer | 10 | 1

BASELINE CHARACTERISTICS:
Population: 158 patients and 158 caregivers participated in this dyadic research. We report age, gender, and ethnicity for total individuals by combining patients and caregivers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Family SWaP Intervention | Usual Care | Total
Number analyzed (Participants) | 158 | 158 | 316
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 98 | 198
  >=65 years | 58 | 60 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 86 | 174
  Male | 70 | 72 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 156 | 156 | 312
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 23 | 52
  White | 125 | 132 | 257
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 158 | 158 | 316

OUTCOME MEASURES:

1. Primary Outcome: Patients' Adherence to Sodium-restricted Diet Assessed by Urinary Sodium Excretion Levels
Description: Baseline: Patient adherence to a sodium-restricted diet was assessed using 24-hour urinary sodium excretion at 3-time points at baseline, 4-months, and 12 months.
Time Frame: Up to 1 year
Population: Of the 158 patient-caregiver dyads (158 patients with heart failure and 158 primary caregivers), we report the primary outcome of patient adherence to the sodium-restricted diet. Of the 158 patients with heart failure, 79 patients were randomly assigned to the Family Sodium Watchers intervention group and another 79 patients were assigned to the usual care group.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Family SWaP Intervention | Usual Care
Number analyzed (Participants) | 79 | 79
mg/day
  Baseline | 4390.2 (2286.1) | 4048.9 (1969.6)
  4-month | 3338.1 (1580.1) | 4402.9 (2214.6)
  12-month | 3523.1 (2173.3) | 3855.3 (1446.6)

2. Secondary Outcome: All Cause Hospitalization/Mortality
Description: Data for all events of hospitalizations and mortality were collected from the baseline to 12 months follow up.
Time Frame: 12 months
Population: Events included death and hospitalization events for participants.
Measure: Number; unit: first event during follow up
Arm/Group | Family SWaP Intervention | Usual Care
Number analyzed (Participants) | 79 | 79
first event during follow up | 23 | 28

ADVERSE EVENTS:
Time Frame: 1 year follow up from the baseline data collection
Description: We reviewed electronic medical records to identify the first event during 1-year follow-up. Adverse events as the first events in this study include death related to cardiovascular health, death with non-cardiac reasons, inpatient hospitalization related to cardiovascular health, and inpatient hospitalization related to non-cardiac reasons.
Arm/Group | Family SWaP Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/158 | 2/158
Serious Adverse Events (participants affected / at risk) | 23/158 | 28/158
Other Adverse Events (participants affected / at risk) | 0/158 | 0/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family SWaP Intervention (N=158) | Usual Care (N=158)
Cardiac Hospitalization (Cardiac disorders) | 15 (15) | 19 (19) — Inpatient hospitalization related to cardiovascular health conditions
Non-cardiac Hospitalization (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) — Inpatient hospitalization related to non-cardiac reasons. We did not collect specific causes of non-cardiac hospitalization.
Cardiac death (Cardiac disorders) | 3 (3) | 1 (1) — Death related to the cardiovascular health condition
Non-cardiac Death (Investigations) | 1 (1) | 1 (1) — Death related to non-cardiac death. We did not collect specific causes of non-cardiac death.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT03560206/Prot_SAP_ICF_000.pdf